CLINICAL TRIAL: NCT01827163
Title: The Feasibility of Paclitaxel With Trastuzumab and Lapatinib in HER2-Positive Early Stage Breast Cancer
Brief Title: Paclitaxel With Trastuzumab and Lapatinib in HER2-Positive Early Stage Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-002
Record Dates: First submitted 2013-04-02; First posted 2013-04-09 (Estimated); Results first posted 2019-12-18 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-01

CONDITIONS: HER2-Positive Early Stage Breast Cancer
Keywords: Paclitaxel; Trastuzumab; Lapatinib; HER2; 13-002
MeSH Terms: interventions — Paclitaxel; Trastuzumab; Lapatinib; pegfilgrastim

ARMS (1):
- Paclitaxel With Trastuzumab and Lapatinib (Experimental): Paclitaxel (T) at 175 mg/m2 q 2 weeks x 4 with filgrastim/pegfilgrastim + trastuzumab (H) + daily oral lapatinib (L), followed by trastuzumab q 3 weeks x 15 doses + daily oral lapatinib (HL). Pegfilgrastim 6mg will be given subcutaneously (SQ) on day # 2 of each paclitaxel administration. Filgrastim may be used in lieu of pegfilgrastim at physician's discretion. Trastuzumab will be administered weekly (4 mg/kg bolus followed by 2 mg/kg weekly) starting with paclitaxel treatment cycle # 1. After 4 cycles of paclitaxel, pts will receive trastuzumab on a q 3 weeks x 15 doses (to complete about one year). The q 3 week trastuzumab may be started from 1-3 weeks after the last dose of paclitaxel. A total of 15 infusions of trastuzumab will be given q 3 weeks after the completion of paclitaxel during the HL phase. Lapatinib will be given orally at 1000 mg daily, starting with paclitaxel during the THL phase & continued for the remaining year during the HL phase for about a year.
  Interventions: Drug: Paclitaxel; Drug: Trastuzumab; Drug: Lapatinib; Drug: Pegfilgrastim

INTERVENTIONS:
Drug: Paclitaxel
Drug: Trastuzumab — The q 3 week trastuzumab may be started at the last dose of paclitaxel infusion or from 1-3 weeks after the last dose of paclitaxel. Trastuzumab may also be administered at a dose of 6mg/kg during the last dose of paclitaxel in the THL phase.
Drug: Lapatinib
Drug: Pegfilgrastim — Pegfilgrastim SQ is given on day # 2 of each paclitaxel cycle and may be dropped at the last paclitaxel infusion. Filgrastim may be used in lieu of pegfilgrastim at the physician's discretion.

SUMMARY:
The purpose of this study is to study a new treatment for HER2-positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed adenocarcinoma with HER2/neu immunohistochemistry 3+ or FISH-amplified breast cancer with a ratio of ≥ 2.0
* Tumor size of ≤ 3 cm and node-negative disease. Nodes with single cells or tumor clusters < 0.2 mm by H&E or IHC are considered node-negative. Patients with micrometastasis (nodes with tumor clusters between 0.02 and 0.2 cm) are allowed. Further axillary dissection will be determined by the patient's surgeon as per standard of care.
* Patients must be ≥18 years of age.
* Patients must have an ECOG performance status of 0 or 1.
* Treatment should be started within 90 days of the final surgical procedure for breast cancer.
* Patients may have bilateral synchronous breast tumors. Patients may have received hormonal therapy for the purpose of chemoprevention but must be willing to discontinue prior to enrollment and while participating in this trial.
* If patients have peripheral neuropathy, it must be ≤ grade 1.
* Patients must be willing to discontinue sex hormonal therapy e.g., birth control pills, ovarian hormonal replacement therapy, etc., prior to enrollment. Women of childbearing potential must be willing to consent to using effective contraception while on treatment and for a reasonable period thereafter.
* Hematologic parameters: absolute neutrophil count (ANC) ≥1500/μL and platelet count ≥100,000/μL.
* Non-hematologic parameters: total bilirubin must be ≤ 1.5 X institutional upper limit of normal (ULN), transaminases (SGOT or SGPT) ≤ 3.0 x ULN.
* Negative HCG pregnancy test for premenopausal women of reproductive capacity and for women less than 12 months after the menopause. LVEF by ECHO (with strain if possible) with LVEF of ≥ 50%. If an ECHO cannot be done, a MUGA may be performed.
* Patients must give written, informed consent indicating their understanding of and willingness to participate in the study.

Exclusion Criteria:

* Patients with stage IV breast cancer or undergoing chemotherapy, radiation therapy, immunotherapy, or biotherapy for current breast cancer.
* Pregnant or breastfeeding patients.
* Patients with a concurrently active second malignancy, other than adequately treated non-melanoma skin cancers or in situ cervical cancer.
* Patients with unstable angina, congestive heart failure, or with a history of a myocardial infarction within 12 months. Patients with high-risk uncontrolled arrhythmias (ventricular tachycardia, high-grade AV block, supraventricular arrhythmias which are not adequately rate-controlled). Patients are excluded if they have grade 3 QT prolongation (Appendix F) (>500 ms) or require drugs that may prolong the QT.
* Subjects who have current active hepatic (including hepatitis B or C) or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones).
* Patients with active, unresolved infections.
* Patients with a sensitivity to E. coli derived proteins.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chau Dang, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan-Kettering Cancer Commack, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Rockville Centre, Rockville Centre, New York

REFERENCES:
- [Derived] Iyengar NM, Fornier MN, Sugarman SM, Theodoulou M, Troso-Sandoval TA, D'Andrea GM, Drullinsky PR, Gajria D, Goldfarb SB, Comen EA, Lake DE, Modi S, Traina TA, Lacouture ME, Chen MF, Patil S, Baselga J, Norton L, Hudis CA, Dang CT. A Pilot Study of Dose-Dense Paclitaxel With Trastuzumab and Lapatinib for Node-negative HER2-Overexpressed Breast Cancer. Clin Breast Cancer. 2016 Apr;16(2):87-94. doi: 10.1016/j.clbc.2015.09.009. Epub 2015 Sep 25. PMID 26454612
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Paclitaxel With Trastuzumab and Lapatinib: Paclitaxel (T) at 175 mg/m2 q 2 weeks x 4 with filgrastim/pegfilgrastim + trastuzumab (H) + daily oral lapatinib (L), followed by trastuzumab q 3 weeks x 15 doses + daily oral lapatinib (HL). Pegfilgrastim 6mg will be given subcutaneously (SQ) on day # 2 of each paclitaxel administration. Filgrastim may be used in lieu of pegfilgrastim at physician's discretion. Trastuzumab will be administered weekly (4 mg/kg bolus followed by 2 mg/kg weekly) starting with paclitaxel treatment cycle # 1. After 4 cycles of paclitaxel, pts will receive trastuzumab on a q 3 weeks x 15 doses (to complete about one year). The q 3 week trastuzumab may be started from 1-3 weeks after the last dose of paclitaxel. A total of 15 infusions of trastuzumab will be given q 3 weeks after the completion of paclitaxel during the HL phase. Lapatinib will be given orally at 1000 mg daily, starting with paclitaxel during the THL phase & continued for the remaining year during the HL phase for about a year.
  Paclitaxel
Period: Overall Study
Arm/Group | Paclitaxel With Trastuzumab and Lapatinib
Started | 20
Completed | 9
Not Completed | 11
Not completed — Hypersensitivity reaction to Paclitaxel | 2
Not completed — Adverse Event | 9

BASELINE CHARACTERISTICS:
Arm/Group | Paclitaxel With Trastuzumab and Lapatinib
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 49 [33 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 16
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Are Able to Complete THL (Paclitaxel, Trastuzumab, and Lapatinib) Without a Dose Delay or Reduction, Grade 3 or Greater QTc Prolongation
Description: The primary objective of this trial is to determine the feasibility of this regimen in patients with node-negative HER-2/neu overexpressed /amplified breast cancer with a tumor size of < 3 cm. The regimen is considered feasible if patients are able to complete the paclitaxel, trastuzumab, and lapatinib (THL) portion of the regimen without a dose delay or reduction or grade 3 or greater QTc prolongation.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Paclitaxel With Trastuzumab and Lapatinib
Number analyzed (Participants) | 20
Participants
  Did not complete treatment | 16
  Successfully completed treatment | 4

2. Secondary Outcome: Participants Toxicity Evaluated While on Study Treatment
Description: All toxicities following chemotherapy will be graded using the National Cancer Institute - Common Toxicity Criteria version 4.0.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Paclitaxel With Trastuzumab and Lapatinib
Number analyzed (Participants) | 20
Participants | 20

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Paclitaxel With Trastuzumab and Lapatinib
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 4/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paclitaxel With Trastuzumab and Lapatinib (N=20)
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Breast infection (Infections and infestations) | 1
Creatinine increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Fatigue (General disorders) | 1
Fever (General disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Hypertension (Vascular disorders) | 1
Transient ischemic attacks (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paclitaxel With Trastuzumab and Lapatinib (N=20)
Diarrhea (Gastrointestinal disorders) | 16
Fatigue (General disorders) | 16
Skin & subcutaneous tissue disorders Other, spec (Skin and subcutaneous tissue disorders) | 16
Peripheral sensory neuropathy (Nervous system disorders) | 12
Alopecia (Skin and subcutaneous tissue disorders) | 11
Rash acneiform (Skin and subcutaneous tissue disorders) | 9
Alanine aminotransferase increased (Investigations) | 8
Bone pain (Musculoskeletal and connective tissue disorders) | 8
Hot flashes (Vascular disorders) | 8
Mucositis oral (Gastrointestinal disorders) | 8
Pain (General disorders) | 8
Anemia (Blood and lymphatic system disorders) | 7
Nausea (Gastrointestinal disorders) | 7
Alkaline phosphatase increased (Investigations) | 6
Dizziness (Nervous system disorders) | 6
Dyspepsia (Gastrointestinal disorders) | 6
Fever (General disorders) | 6
Irregular menstruation (Reproductive system and breast disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Aspartate aminotransferase increased (Investigations) | 4
Constipation (Gastrointestinal disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 4
Musculoskeletal & conn tissue disorder Other, spec (Musculoskeletal and connective tissue disorders) | 4
Anorexia (Metabolism and nutrition disorders) | 3
Blood bilirubin increased (Investigations) | 3
Chills (General disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Edema limbs (General disorders) | 3
Headache (Nervous system disorders) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 3
Memory impairment (Nervous system disorders) | 3
Nervous system disorders - Other, specify (Nervous system disorders) | 3
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
Weight loss (Investigations) | 3
Dehydration (Metabolism and nutrition disorders) | 2
Dry eye (Eye disorders) | 2
Dysgeusia (Nervous system disorders) | 2
Dysphagia (Gastrointestinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypertension (Vascular disorders) | 2
Hypoglycemia (Metabolism and nutrition disorders) | 2
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 2
Nail loss (Skin and subcutaneous tissue disorders) | 2
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2
Urinary frequency (Renal and urinary disorders) | 2
Vaginal dryness (Reproductive system and breast disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
White blood cell decreased (Investigations) | 2
Allergic reaction (Immune system disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Anal hemorrhage (Gastrointestinal disorders) | 1
Anxiety (Psychiatric disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Ataxia (Nervous system disorders) | 1
Blurred vision (Eye disorders) | 1
Breast pain (Reproductive system and breast disorders) | 1
Conjunctivitis (Eye disorders) | 1
Creatinine increased (Investigations) | 1
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
INR increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Metabolism and nutrition disorders-Other (Metabolism and nutrition disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Nail infection (Infections and infestations) | 1
Nail ridging (Skin and subcutaneous tissue disorders) | 1
Paronychia (Infections and infestations) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1
Rash pustular (Infections and infestations) | 1
Renal and urinary disorders - Other (Renal and urinary disorders) | 1
Resp, thoracic & mediastinal disorder - Other (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis infective (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Transient ischemic attacks (Nervous system disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Watering eyes (Eye disorders) | 1
Weight gain (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-28): https://cdn.clinicaltrials.gov/large-docs/63/NCT01827163/Prot_SAP_000.pdf